CLINICAL TRIAL: NCT00517998
Title: Phase 1 Study of the Biologic Lung Volume Reduction (BLVR) System in Patients With Advanced Emphysema
Brief Title: Israeli Biologic Lung Volume Reduction (BLVR) Phase 1 Emphysema Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Edward P Ingenito, MD, PhD, Medical Director & CSO, Aeris Therapeutics Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-C06-002
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Pulmonary Emphysema; Chronic Obstructive Pulmonary Disease
Keywords: Lung volume reduction; Bronchoscopy; Emphysema; COPD; NETT; Lung disease; COLD; BLVR
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Emphysema; Lung Diseases | interventions — Hydrogels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group1 (Experimental): Treatment will be administered in two sessions.
  Interventions: Drug: Biologic Lung Volume Reduction (BLVR) - 10 mL Hydrogel
- Group2 (Experimental): Treatment will be administered in a single session.
  Interventions: Drug: Biologic Lung Volume Reduction (BLVR) - 10 mL Hydrogel

INTERVENTIONS:
Drug: Biologic Lung Volume Reduction (BLVR) - 10 mL Hydrogel — 10 mL Hydrogel

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Biologic Lung Volume Reduction System (BLVR) for patients with advanced emphysema refractory to medical therapy.

DETAILED DESCRIPTION:
Background:

Patients with emphysema currently have limited treatment choices. Many patients are treated with steroids and inhaled medications, which often provide little or no benefit. In recent years, lung volume reduction surgery has become an accepted therapy for advanced emphysema. Lung volume reduction surgery involves the removal of diseased portions of the lung in order to enable the remaining, healthier portions of the lung to function better. This procedure, although effective for many patients, is complicated and is accompanied by substantial morbidity and mortality risk.

Aeris Therapeutics has developed the Biologic Lung Volume Reduction (BLVR) System which is intended to achieve lung volume reduction without surgery and its attendant risks. Patients are treated using a bronchoscope to direct treatment to the most damaged areas of the lung. The treatment delivers a precisely proportioned proprietary mixture of drugs and biologics which, when combined at the treatment site, form a biodegradable hydrogel. The hydrogel acts to reduce lung volume by permanently collapsing and sealing the diseased areas of the lung. This provides room within the chest to allow the remaining healthier portions of the lung to function better.

Aeris' BLVR development program has been granted Fast Track designation by the U.S. FDA, and is the subject of ongoing clinical trials designed to investigate the safety and efficacy of the BLVR System as a treatment for patients with advanced heterogeneous emphysema. Fast Track designation is reserved for drug and biologic development programs that are intended to treat serious or life-threatening conditions and that demonstrate the potential to address unmet medical needs.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of advanced emphysema
* age >/= 40 years
* clinically significant dyspnea
* failure of standard medical therapy to relieve symptoms (inhaled beta agonist & inhaled anticholinergic)
* pulmonary function tests within protocol-specified ranges (post bronchodilator FEV1 < 45% predicted & experiencing < 30% or 300 mL improvement using bronchodilator; total lung capacity > 110% predicted; residual volume > 150% predicted)
* 6 Minute Walk Distance >/= 150 m

Exclusion Criteria:

* alpha-1 protease inhibitor deficiency
* tobacco use within 4 months of initial visit
* body mass index < 15 kg/m2 or> 35 kg/m2
* clinically significant asthma, chronic bronchitis or bronchiectasis
* allergy or sensitivity to procedural components
* pregnant, lactating or unwilling to use birth control if required
* prior lung volume reduction surgery, lobectomy, pneumonectomy, lung transplant, endotracheal valve placement, airway stent placement or pleurodesis
* comorbid condition that could adversely influence outcomes
* significant comorbidity

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
SAEs - Safety of treatment and the procedure | 1 year

SECONDARY OUTCOMES:
Reduction in gas trapping | 12 weeks
Improvement in exercise capacity | 12 weeks
Improvement in lung function (vital capacity) | 12 weeks
Improvement in lung function (expiratory flow) | 12 weeks
Improvement on dyspnea symptoms | 12 weeks
Improvement in quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yael Refaely, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tivka, Israel

REFERENCES:
- [Background] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835
- [Background] Reilly J, Washko G, Pinto-Plata V, Velez E, Kenney L, Berger R, Celli B. Biological lung volume reduction: a new bronchoscopic therapy for advanced emphysema. Chest. 2007 Apr;131(4):1108-13. doi: 10.1378/chest.06-1754. PMID 17426216